# Statistical Analysis Plan

| Sponsor | |
|---|---|
| Protocol Title: | A Prospective, Randomized, Blinded Evaluator, Multicenter, Between-subjects Clinical Study to Evaluate Safety and Effectiveness of RHA® 4 versus for Treatment of Midface Volume Deficiency |
| Protocol Number: | |
| Document Version: | |
| Document Date: | 21-Jul-2023 |

# **Approvals**

| Role | Signatures |
|-----------------|-------------|
| | Print Name: |
| | Cian Nama |
| | Sign Name: |
| Biostatistician | |
| | Print Name: |
| | Sign Name: |
| Peer Reviewer | |

AD-ST-33.06 Effective date: 12-Nov-2020



# **Document History**

| Version | Date | Author | Description |
|---------|------|--------|-------------|



# **List of Abbreviations**

| Abbreviation | Definition |
|--------------|-------------------------------------------|
| ADE | Adverse Device Effect |
| AE | Adverse Event |
| BLE | Blinded Live Evaluator |
| BMI | body mass index |
| CI | Confidence Interval |
| CIP | Clinical Investigation Plan |
| COVID-19 | Coronavirus Disease 2019 |
| CSR | Clinical Study Report |
| CTR | Common Treatment Response |
| eCRF | electronical Case Report Form |
| FDA | Food and Drug Administration |
| GAIS | Global Aesthetic Improvement Scale |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |

| Abbreviation | Definition |
|--------------|-------------------------------------------|
| UPT | Urine Pregnancy Test |
| US | United States |
| WHO-DD | world health organization drug dictionary |

| Statistic | al Ana | lysis P | an |
|-----------|--------|---------|----|
| Protoco | Numl | per | |

| 1.2. | Hypothesis |
|---|---|
| midfac | HA4 group will be statistically non-inferior to the group for the treatment of see volume deficiency as determined by the Teoxane Midface Volume Deficit Scale DS – 5-point scale 8 weeks after the last treatment (initial or touch-up). |
| A char<br>meanii | nge in the TMVDS ≥1 grade compared to pretreatment will be considered clinically ngful. |
| 2. | Study Objectives and Endpoints |
| 2.1. | Study Objectives |
| The st | udy is designed to achieve a series of objectives outlined below. |
| 2.1.1. | Primary Effectiveness Objective |
| midfac | ess the effectiveness (non-inferiority) of RHA4 versus on adding volume in the ce region in subjects seeking treatment of midface volume deficiency 8 weeks after the last ent (initial or touch-up). |
| 2.1.2. | Secondary Effectiveness Objectives |
| The se | condary objectives are: |
| • | To assess the effectiveness of RHA4 versus on adding volume in the midface region in subjects seeking treatment of midface volume deficiency up to 52 weeks after last treatment and 12 weeks after retreatment |
| 2.1.3. | Safety Objective |
| i <b>⊕</b> 9 | To assess the safety of RHA4 versus in subjects undergoing treatment of midface volume deficiency up to 52 weeks after last treatment and 12 weeks after retreatment |
| 10 | |





### 2.2.2. Safety Endpoints

The safety endpoints of this study include the following:

 Adverse events (AEs) with a focus on treatment related AEs based on the TI assessment, and AEs reported from the Common Treatment Response (CTR) diary



Each AE will be coded to a Preferred Term (PT) and associated System Organ Class (SOC) according to an established and validated adverse reaction dictionary (Medical Dictionary for Regulatory Activities [MedDRA], latest available version) before the randomized treatment code

| At Screening (Visit 0), the TI will evaluate the subject's midface using the 5-grade Teoxane Midface Volume Deficit Scale (TMVDS) for eligibility of the subject |
|---|
| The BLE will evaluate the subject's midface using the TMVDS at Screening to confirm eligibility. This will be done independently of the TI. If the assessments of the TI and the BLE are the same or differ exactly by 1 point of the scale, the difference will be considered acceptable. |
| Subjects who are eligible to participate in the main study will be enrolled and randomly assigned in a 3:1 ratio to receive RHA4 or |
| Administration and Evaluation |
| At Visit 1, continuous eligibility will be assessed. All evaluations performed at Visit 1 before the injection will be considered for the Baseline. |
| The TI will inject the device at Visit 1. |
| Administration of will follow the instructions for use (IFU), the TI can use an FDA-approved needle and/or cannula as per their choice, at each injection. |
| RHA4 can be injected with a needle, and/or with a cannula; this will be left to the choice of the |




The primary endpoint of the study is the difference in the TMVDS change from Baseline to 8 weeks after the last day of treatment between subjects treated with RHA4 and those treated with mith.

A Per Protocol (PP) and Intent-to-treat (ITT) analysis sets will be used for the effectiveness analysis.



The devices used for administration must be approved for the use by the US FDA.

<u>Injection area</u>: The TEOXANE SA midface treatment area will focus on the anteromedial and lateral malar regions. The treatment area is delimited using the following triangle: its base line is parallel to the nasolabial fold (at least 0.4" [1 cm] lateral to the fold), the superior side of the triangle is a line from the superior part of the nasal alar crease to the superior root of the helix of the ear and the inferior side of the triangle is a line running from the lateral oral commissure to the superior root of the helix of the ear.

Treatment of nasolabial folds, temples, pre-auricular and periorbital regions are prohibited.

Amount of device to administer: The maximum volume per administration of RHA4 and into the midface area is 6.0 mL per treatment session (total for both sides of the face, i.e., 3.0 mL maximum per side).

# 3.5. Method of Assigning Subjects to Treatment Groups

The randomization schedule will be computer generated using a permuted block algorithm and randomly allocate the investigational product in a 3:1 ratio. Subject will be randomized to one of the following groups:

- RHA® 4 study device
- control device.



#### 3.6. Blinding and Unblinding

The TI, unblinded to treatment allocation, will be asked to minimize the number of people who will have treatment allocation information or who will have any form of access to such information. Access will only be given to personnel who must have it to, for example, administer the filler, call the subjects, or schedule visits.

The BLE and study personnel not involved with the site (e.g., data management, medical monitor) will be blinded to treatment assignment. All evaluations performed by the BLE will be









#### 6.1.6.5. Prior and Concomitant Medications

Medications that started prior to the initial treatment will be considered prior medications.

A concomitant medication is defined as any medication that was administered during the treatment period. This includes medications that started before the treatment period and continued while on treatment and medications that started during the treatment period.

If the start/stop dates of a medication are partially or completely missing, then the medication will be assumed to be concomitant if it cannot be definitely shown that it was not administered during the treatment period. Missing dates will not be replaced.

### 6.1.7. Data Adjustments/Handling/Conventions

All collected data will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included only in the data listings.

Subjects retreated with an unexpected treatment at Visit 7 will have their assessments performed after retreatment excluded from the analysis and only listed.

All P values will be displayed in 4 decimals and rounded using standard scientific notation (eg, 0.XXXX). If a P value less than 0.0001 occurs it will be shown in tables as < 0.0001.

For missing AEs onset dates, the convention for replacing missing dates for the purposes of calculating derived variables is as follows:

For partial AE start dates:

- If the year is unknown, then do not impute the date but assign a missing value.
- If the month and day are unknown, then:
  - o If the year matches the year of injection date, and the end date (if present) is after injection date, then impute as the month and day of the injection date.
  - o Otherwise, assign January.
- If the month only is unknown, then:
  - o If the year matches the year of injection date and day is on or after day of injection, then assign the month of injection. If this produces a date after the AE end date, assign the month before.
  - o If the year matches the year of injection date and day is before day of injection, then assign the month after injection. If this produces a date after the AE end date, assign the month of injection.
  - Otherwise, assign January.
- If the day is unknown, then:
  - o If the month and year match the month and year of the injection date, then impute as the day of injection date. If this produces a date after the AE end date, assign 01.
  - o Otherwise, assign 01.

For partial AE end dates:

All protocol deviations will be listed.

# 7.3. Demographics and Other Baseline Characteristics

Descriptive summaries of the <u>demographics</u> (age, sex, height, body weight, calculate body mass index (BMI), ethnicity, race, Fitzpatrick skin type) will be completed for each of the following populations: ITT, Safety and PP.

For the continuous variables, the number of non-missing values and the mean, SD, minimum, median and maximum will be tabulated.

Descriptive summaries of the <u>medical/surgical history and prior medications</u> will be completed for the Safety population.

Medical/surgical history will be coded with MedDRA dictionary. Incidences of findings in medical history will be summarized by SOC and PT, unless otherwise specified.

The frequency and percentage of prior medications will be summarized using the latest version available at time of the database lock of the World Health Organization Drug Dictionary (WHO-DD) by Anatomical Therapeutic Chemical (ATC) level 2 within level 1.

#### 7.4. Exposure and Compliance

Data will be tabulated for Safety population.

Number of treatment sessions will be tabulated in a frequency table by treatment group.

Total volume to obtain an OCR (initial treatment and touch-up summed) and volume injected at each treatment session will be tabulated in a summary table by treatment group.

Method of administration, injection technique, depth of injection where device was injected will be tabulated in a frequency table by treatment group.

Number of device malfunction reported by visit will be tabulated in a frequency table by treatment group.

All exposure data will be listed.

#### 8. Effectiveness Analysis




Statistical Analysis Plan



The following categories are used:

- Responder
- Non-responder





## 8.2.5. Subject Satisfaction Score

Subject Satisfaction will be assessed by subjects using the following static 5-grade scale. Grade description:

1. Very satisfied



#### 5. Very dissatisfied.

Satisfaction grade frequencies and percentages will be calculated and presented for each scheduled study visit by treatment arm.

For subject satisfaction, proportions of "satisfied" and "very satisfied" (subject satisfaction responder rate) will be presented, along with the 95% CI of the proportion at each applicable study visit.





Adverse events will be recorded either directly by the TI or will come from CTR diary per thei duration

All AEs reported during the study will be described by SOC and PT.

Incidence rates defined as number of subjects presenting the AE divided by the number of subjects in the treatment group with 2-sided exact 95% CIs will be calculated for the overall incidence of AEs, ADEs,

The causal relationship of the AE to the study treatment is determined by the investigator by relationship to the study procedure and relationship to the study device

# 9.1.1. Deaths and Serious Adverse Events

All deaths occurring during the study will be listed.

All SAEs occurring during the study will be listed.

#### 9.2. CTRs

Number of all CTRs and number and percentage of subjects having the specific CTR will be presented for each injection.

CTRs to be reported are the following;

- o Redness
- o Pain
- Tenderness
- o Firmness
- o Swelling
- o Lumps/Bumps
- o Bruising
- o Itching
- o Discoloration





# 10. COVID-19 Impact

Visits and assessments impacted by the COVID-19 pandemic will be listed.









Statistical Analysis Plan

Protocol Number



# 15. Tables, Listings, and Listing Shells

# 15.1. Standard Layout for all Tables, Listings, and Figures

The following standard layout will be applied to all Tables, Listings, and Figures in support of this study. Note that programming notes may be added if appropriate after each tables, listings and figures (TLF) shell.



# 15.2. Planned Table Shells

Will be provided in separate document.



# 15.4. Planned Figure Shells

Will be provided in separate document.







**Appendix 2: Clinical Investigation Design** 

